CLINICAL TRIAL: NCT01877707
Title: A Home-based, Rapid and Quantitative Test for Bacterial Respiratory Infections in Patients With Cystic Fibrosis, to Reduce Admissions and Hospital Stay Length and to Improve Healthcare Outcomes.
Brief Title: Near Patient Microbial Testing in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Judy Ryan, Research & Database Manager, Papworth Hospital NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12/EE/0462
Record Dates: First submitted 2013-06-07; First posted 2013-06-14 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cystic Fibrosis patients (Other): Patients with a diagnosis of cystic fibrosis, who are able to produce daily sputum samples. With a history of at least two pulmonary infective exacerbations within the past 12 months.
  Interventions: Other: home monitoring

INTERVENTIONS:
Other: home monitoring — Record daily - peak flow measurements, pulse rate, oxygen saturation levels, weight,activity and daily sputum samples.

SUMMARY:
To identify whether home monitoring of multiple physiological parameters and biomarkers in sputum could provide advanced warning of an infective exacerbation or treatment failure before changes in patient-reported symptoms.

DETAILED DESCRIPTION:
1. To determine if longitudinal profiling of sputum from Cystic Fibrosis patients allow accurate prediction of exacerbations in a study of a larger group and can we confirm the 7+ day early warning system works in this larger group.
2. Is one biomarker sufficient to predict exacerbations - what is the accuracy? Are two or more biomarkers required to achieve an accuracy of greater than 95%?
3. Can we now accurately determine how many hospital bed days a home testing/wellness monitoring device would save? What is the business case for healthcare providers to adopt our future test for home use? We estimate a 50% saving. Can this be confirmed?
4. When used in the clinic, how many hospital days would our test save through faster determination of treatment efficacy? What is the business case for adopting our future test as a point of care test on the ward in Cystic Fibrosis centres? Could this be the new revolutionary tool that we anticipate?
5. We forecast a 50% reduction in costs to treat Cystic Fibrosis patients in disease severity bands 2-A to 5. Can we provide evidence for this to support further investment?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis based on genetic testing and/or sweat chloride levels.
* Chronic infection with Pseudomonas aeruginosa.
* Patients able to produce daily sputum samples.
* Current history of at least two pulmonary infective exacerbations in the past 12 months.
* Able to give written informed consent

Exclusion Criteria:

* Unable to provide written informed consent
* Patients unable to produce daily sputum samples
* Fewer than two infective pulmonary exacerbations in 12 months

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Advance warning of an infective exacerbation | one year
  To identify whether home monitoring of multiple physiological parameters and biomarkers in sputum could provide advanced warning of an infective exacerbation or treatment failure before changes in patient-reported symptoms.
  Participants will collect daily sputum samples which will be profiled for psuedomonas aeruginosa.

SECONDARY OUTCOMES:
home monitoring of multiple physiological parameters | one year
  1. Daily peak flow measurements will be obtained for FEV1 and PEF
  2. Daily pulse rate and oxygen saturations levels
  3. Participants will weigh themselves daily on study specfic scales
  4. Participants will wear a step counter during waking hours to measure their activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Floto, MA, MRCP, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Trust, Cambridge, United Kingdom